CLINICAL TRIAL: NCT02731560
Title: Efficacy and Safety of Rituximab in Pakistani Patients With Rheumatoid Arthritis (RA)
Brief Title: Rituximab (RTX) for Disease Modifying Anti Rheumatic Drug (DMARD) Non-responders in Pakistan: The Pakistan Rituximab Study (PARIS)
Acronym: PARIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Abid Z. Farooqi (Other Government)
Collaborators: Aga Khan University (Other); Fatima Memorial Hospital (Other); Fauji Foundation Hospital (Other)
Responsible Party: Sponsor-Investigator, Prof. Abid Z. Farooqi, Professor of Rheumatology, Pakistan Institute of Medical Sciences
Organization: Pakistan Institute of Medical Sciences (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25190
Record Dates: First submitted 2016-03-06; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Pakistan, Rituximab; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Treatment with Rituximab in RA patients showing inadequate response to standard DMARDs
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab was administered as an intravenous infusion as per approved protocol on Day 1 and day 14. The protocol stipulated the administration of intravenous hydrocortisone 100 mg and oral pheniramine maleate 43.5 mg as pre-medication. The Rituximab itself was given as a 1 gm infusion slowly over a period of 4-6 hours.
  This was done either by a specialist nurse or a trained doctor.
  Other Names: RTX

SUMMARY:
A study to determine the efficacy and safety of rituximab in Pakistani patients with rheumatoid arthritis (RA) who have been inadequately controlled with standard disease modifying anti rheumatic drugs (DMARDs).

DETAILED DESCRIPTION:
Enrolled subjects with inadequately-controlled RA had their disease activity level assessed before initiation of therapy and at intervals of 6 months and 12 months thereafter. Standardized disease activity scores like the Disease Activity Score-28 (DAS 28) were used for determining remission or otherwise of the disease. The American College of Rheumatology (ACR) 20, 50 and 70 response scores and the European League of Associations for Rheumatology (EULAR) Response Criteria for RA were used to determine the percentage improvement in the individual subject's condition at the same intervals. The former utilizes a set of assessments to determine if, after a given therapy, there has been a 20, 50 or 70% improvement in the aggregate scores as compared to the baseline and the latter utilizes calculated improvements in the DAS 28 score to determine if the response to treatment has been good, moderate or none. Both of these have been validated and approved for use by the ACR and EULAR respectively.

The study enrollment period was from 1st January 2010 till 31st December 2010. Observation period was 12 months from the enrollment date for each subject. The final results are being reported here.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Men and women aged 18-80 years, inclusive.
3. Patients with RA for at least 6 months.
4. DAS28 score > 3.70 at baseline.
5. Inadequate response to methotrexate (MTX), for at least 4 weeks using a stable dose of 15mg/week. Glucocorticoids (<10 mg/day prednisone or equivalent) permitted if stable for at least 4 weeks prior to baseline.
6. Use of Non-steroidal anti-inflammatory drugs (NSAIDs) permitted if stable dose for at least 2 weeks prior to baseline.
7. Patients of reproductive potential (males and females) must be willing to use a reliable method of contraception (e.g. contraceptive pill, intrauterine device (IUD) or a physical barrier) during the study and for 12 months after last Rituximab administration.
8. If female and of childbearing potential, a negative serum pregnancy test within 2 weeks prior to baseline.

Exclusion Criteria:

Exclusion Criteria Related to RA

1. Bed bound or wheelchair bound patients.
2. Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA

Exclusions Related to Medications

1. History of severe allergic or anaphylactic reactions to a biologic agent or known hypersensitivity to any component of Rituximab or to murine proteins.
2. Previous treatment with any approved or investigational biologic agent for RA.
3. Concurrent treatment with any biologic agent for any indication.
4. Receipt of any vaccine within 4 weeks prior to baseline (it was recommended that a patient's vaccination record and the need for immunization prior to receiving Rituximab should be carefully investigated).
5. Intolerance to or contraindications to drugs required for the treatment of adverse event of Rituximab (e.g., paracetamol, anti-histamines, hydrocortisone, anti-emetics or histamine-receptor 1 (H1) blockers).
6. Intra-articular or parenteral glucocorticoids within 4 weeks prior to baseline.

Exclusions for General Safety/Health

1. Any surgical procedure, including bone / joint surgery / synovectomy (including joint fusion or replacement) within 12 weeks prior to baseline or planned within 24 weeks of randomization.
2. Evidence of any severe or significant medical condition(s) or disease(s) that, in the view of the investigator, prohibited participation in the study.
3. Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine or gastrointestinal disorders which, in the investigator's opinion, would have precluded patient participation.
4. Significant cardiac (heart failure of New York Heart Association (NYHA) class IV) or pulmonary disease (including obstructive pulmonary disease).
5. Known active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections), or a known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) anti-infectives within 4 weeks prior to baseline or completion of oral anti-infectives within 2 weeks prior to baseline.
6. History of serious recurrent or chronic infection. (for screening for a chest infection a chest radiograph will be performed at screening if not performed within 12 weeks prior to screening).
7. Primary or secondary immunodeficiency (history of, or currently active), including known history of human immunodeficiency (HIV) infection.
8. Pregnancy or breast feeding.
9. Known history of active cancer during the past 5 years, including solid tumours, hematological malignancies and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been excised and cured).
10. Currently active alcohol or drug abuse or history of alcohol or drug abuse within 24 weeks prior to baseline.

Exclusion criteria related to laboratory findings:

1. Positive serum human chorionic gonadotropin measured within two weeks prior to the first infusion of study drug
2. Positive test for hepatitis B surface antigen (HBsAg) or for hepatitis C serology
3. Positive hepatitis B core antibody (HBcAb) associated with positive hepatitis B virus (HBV) detection (> 29 IU/L or > 169 copies/mL)
4. Hemoglobin < 8.0 g/dL
5. Absolute neutrophil count < 1.5 × 103/μL
6. Concentration of serum immunoglobulin G (IgG) and/or immunoglobulin M (IgM) below 5.0 and 0.40 mg/mL, respectively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Disease Activity Assessment Score (DAS-28) | 6 months
  To determine the percentage of previously inadequately-controlled RA patients achieving improvement in their disease activity level post treatment with Rituximab at 6 months interval using Disease Activity Score in 28 selected joints (DAS-28).

SECONDARY OUTCOMES:
Status of disease activity level using DAS 28 score | 12 months
  To determine the percentage of such RA patients achieving improvement in their disease activity level post treatment at 12 months interval using DAS-28.
Status of disease response to treatment using the ACR 20/50/70 response criteria | 12 months
  Using the ACR 20/50/70 response criteria
Status of disease response to treatment using the EULAR response criteria | 12 months
  using the EULAR response criteria
Documenting serious adverse events during the trial period | 12 months
  Any event leading to hospitalization or death during the trial period

CONTACTS AND LOCATIONS:
Overall Officials: Abid Z Farooqi, FRCPI, Principal Investigator — Pakistan Institute of Medical Sciences

IPD SHARING:
Plan to Share IPD: No